CLINICAL TRIAL: NCT06609941
Title: Additive Effects of Alternative Nostril Breathing with Pharmacological Management on Dyspnea and Control Pause in Patients with Bronchial Asthma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/25
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-08

CONDITIONS: Bronchial Asthma
Keywords: Dyspnea, asthma control, peak expiratory flow rate
MeSH Terms: conditions — Asthma; Dyspnea

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial having two groups. One group will receive (interventional group) alternative nostril breathing along with pharmacological management and the other group (control group) will receive only pharmacological management.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nostril Breathing along with pharmacological therapy Group (Experimental): Patients in this group will receive alternative nostril breathing along with pharmacological management.
  Total 4 weeks protocol. Two sessions per week will be supervised by physiotherapist and 5 days at home. A home diary will be provided in order to ensure and follow-up that participants are performing breathing exercise at home.
  Interventions: Other: Alternative nostril breathing; Drug: Pharmacological therapy
- Pharmacological therapy Group (Active Comparator): Patients will receive medication as prescribed by pulmonologist through stepwise approach according to symptoms and severity. Total 4 weeks protocol.
  Before and after 4 weeks pre and post interventional values will be taken.
  Interventions: Drug: Pharmacological therapy

INTERVENTIONS:
Other: Alternative nostril breathing — Patients in this group will receive alternative nostril breathing along with pharmacological management. For alternative nostirl breathing patient will be advised to inhale slowly (4sec) and deeply through left nostril.Then hold breath for 2-3 sec. Release right nostril and use right ring finger to close left nostril. Exhale slowly (6sec) and completely through right nostril. Inhale slowly (4sec) and deeply through right nostril. Then hold breath for 2-3sec. Release left nostril and use right thumb to close right nostril. Exhale slowly (6sec) and completely through left nostril. Repeat the cycle.
  Arms: Nostril Breathing along with pharmacological therapy Group
Drug: Pharmacological therapy — Participants in this group will only be provided with standard pharmacological management for 4 weeks as prescribed by a pulmonologist. For example:
  Salbutamol inhaler (Short acting bronchodilator) Saltra inhaler (Selective long acting β2 adrenoceptor agonist) Tiotropium (Anticholinergic) Combivir (Nucleoside analogue - reverse transcriptase inhibitor) etc.
  Week 01 and week 02:
  Patients will receive medication prescribed by pulmonologist.
  Week 03 and week 04:
  Patients will receive medication prescribed by pulmonologist.

SUMMARY:
Bronchial asthma is a widespread chronic condition charactrized by inflammation and narrowing of airways, leading to repeateted episodes of breathlessness, wheezing and labored breathing.Breathing exercises help to manage hyperventilation often seen in asthmatic patients. To handle respiratory complications asthmatics are advised to practise nasal breathing techniques in conjunction with their prescribed medications.

DETAILED DESCRIPTION:
Bronchial asthma is a very common chronic disease marked by inflammation and constriction of airways, resulting in recurrent episodes of breathlessness, wheezing and decrease work of breathing. Breathing exercises help to manage hyperventilation associated with asthma. In order to manage respiratory conditions asthmatic patients are encouraged for nasal breathing techniques along with pharmacological management. Hence the objective of the study is to compare the effects of alternative nostril breathing along with pharmacological management versus pharmacological management alone on dyspnea, control pause, asthma control and peak expiratory flow rate in patients with bronchial asthma.

ELIGIBILITY:
Inclusion Criteria:

* Adults: aged (18-45 years)
* Gender: Both males and females
* Grade1- Grade 4 on Modified MRC dyspnea scale
* Asthma severity classes (intermediate, mild persistent and moderate persistent asthma) acc. to NAEPP national asthma education and prevention program guidlin

Exclusion Criteria:

* Patients having acute exacerbation of COPD or status asthmaticus
* Patients diagnosed with acute infections
* Patients unable to follow command/ instructions
* Asthma patients with >40 sec control pause duration
* Patients who fall in red zone of asthma action plan (PEFR < 50%)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Dyspnea | 4 weeks
  Evaluation will be done using Dyspnea-12 questionnaire for dyspnea
Control pause | 4 weeks
  Stopwatch will be used to measure control pause.
Asthma control | 4 weeks
  Asthma control test (ACT) will be used to evaluate asthma control and peak flow meter for peak expiratory flow rate.
Peak expiratory flow rate. | 4 Weeks
  Peak flow meter will be used to measure peak expiratory flow rate

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan